CLINICAL TRIAL: NCT04204590
Title: Feasibility Study of a Systematic Approach for Deprescribing of Statins and Proton Pump Inhibitors in Nursing Home Residents
Brief Title: Feasibility Study of a Systematic Approach for Deprescribing of Statins and PPI's.
Acronym: FeDeS+P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z2018001
Record Dates: First submitted 2018-05-01; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Polypharmacy
Keywords: Deprescribing

STUDY DESIGN:
Intervention Model Description: A multicentre, unblinded, single group (pre-comparison and post-comparison) feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): The aim of this study is to test the feasibility of this algorithm as an intervention to carry out deprescribing a targeted medication group, proton pump inhibitors (PPI's) and statins, among nursing home residents.
  Interventions: Other: Deprescribing algorithm

INTERVENTIONS:
Other: Deprescribing algorithm — For this study an implicit, evidence-supported and patient-centred algorithm has been developed. The outcome of the algorithm is an advice to the doctor to deprescribe or not deprescribe the statin and/or PPI.

SUMMARY:
Deprescribing, the process of safely reducing or discontinuing unnecessary or harmful medication, has the potential to decrease polypharmacy and improve health outcomes. In this study a structured implicit algorithm, focusing on both extrinsic medication factors (eg change in disease) and intrinsic patient factors (eg. pill burden) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participant uses a statin and/or a proton pump inhibitor.
* Participant signs informed consent.
* Participant is a nursing home resident.

Exclusion Criteria:

* Participant is there for short term nursing home admission (<3 months)
* Participant is there for hospice admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Decrease in pill burden (the number of statins and PPI's) | 3 and 6 months after intervention.
  On T0 (intervention) and on T1 + T2 (3 and 6 months after intervention), we will measure the number of PPI's and statins on the medication list of every participant. These are provided by the pharmacist.
Decrease in pill burden (the dose of statins and PPI's) | 3 and 6 months after intervention.
  On T0 (intervention) and on T1 + T2 (3 and 6 months after intervention), we will measure the dose of PPI's and statins on the medication list of every participant. These are provided by the pharmacist.

SECONDARY OUTCOMES:
All possible negative side effects of deprescribing (e.g. nausea, symptom recurrence) | From intervention to six months after intervention
  All possible negative effects of deprescribing as recognised by the doctor involved, e.g. symptom recurrence.
Feasibility to use this algorithm. | 3 and 6 months after intervention
  Three and six months after intervention we will ask the participating doctors the next questions (per included participant):
  * What did the algorithm advice you?
  * Did you follow the advice?
  * Why dit you follow/deny the advice?

CONTACTS AND LOCATIONS:
Overall Officials: Jos Schols, Prof. Dr., Principal Investigator — Principal Investigator
Locations (1):
- Lemborgh, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No